CLINICAL TRIAL: NCT05439161
Title: Multicentric Evaluation of Best Corrected Visual Acuity of the XEN Implant Versus Classic Trabeculectomy in Open Angle Glaucoma Subjects
Brief Title: XEN Glaucoma Gel Stent Versus Trabeculectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Dr. Herbert Reitsamer (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. Herbert Reitsamer, Prof. Dr. Herbert Reitsamer, Paracelsus Medical University
Organization: Paracelsus Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A.08242018-v2.15122021
Record Dates: First submitted 2022-06-15; First posted 2022-06-30 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Primary Open Angle Glaucoma; Pseudoexfoliation Glaucoma; Pigmentary Dispersion Glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle; Exfoliation Syndrome | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- XEN Glaucoma Gel Microstent (AbbVie) Device (Active Comparator): Implantation of XEN Glaucoma Gel Microstent (Device, AbbVie) for the treatment of glaucoma will be performed in this arm. It is a newer filtering glaucoma surgery. XEN Glaucoma Gel Microstent implantation accounts to the filtering glaucoma surgeries.
  Interventions: Device: surgery
- Trabeculectomy (Active Comparator): Trabeculectomy will be performed in this arm. Trabeculecomy is the classic filtering glaucoma surgery since more than 50 years for the treatment of glaucoma (gold standard within the filtering glaucoma surgery group).
  Interventions: Device: surgery

INTERVENTIONS:
Device: surgery — 2 types of filtering glaucoma surgeries (classic trabeculectomy as gold standard, and newer XEN glaucoma microstent) are compared against each other in a prospective multicentric randomized study

SUMMARY:
Multicentric evaluation of best corrected visual acuity of the XEN implant versus classic trabeculectomy in open angle glaucoma subjects

DETAILED DESCRIPTION:
The objective of this study is to evaluate the postoperative best corrected visual acuity and refraction in 2 different filtering glaucoma surgeries: XEN implant standalone procedure versus classic trabeculectomy standalone procedure. Both procedures are standard of care in surgical treatment of glaucoma. The XEN implant is a minimally invasive procedure and spares out the dissection of the conjunctiva, while the classic trabeculectomy is a procedure ab externo and supposed to be more invasive.

Up to 196 eyes will be enrolled in both surgery groups. Patients have to be legible for both procedures and are randomly allocated to both groups. Patients, who need a combined cataract procedure are not legible.

A prospective, randomized, multicenter trial. Four study centers in Europe (Austria) will participate.

Patients with open angle glaucoma will be screened for eligibility, and informed consent will be obtained from those who meet screening criteria and are interested in participating in the study. Eligible patients will be examined preoperatively to obtain a medical history and to establish a baseline for the ocular condition. During screening it will be determined via randomization if the subject will be included in group 1 where the XEN implant will be implanted in a standalone procedure or in group 2 where the trabeculectomy will be performed in a standalone procedure. Regardless of study group, all eligible patients will have the same inclusion/exclusion criteria, effectiveness endpoints and follow up exams. An inclusion of both eyes of the same patient is not possible.

Postoperatively, subjects will undergo ophthalmic evaluations at regular intervals as specified in this protocol.

The objective of this study is to evaluate the postoperative best corrected distance and near visual acuity and refraction in 2 different filtering glaucoma surgeries: XEN Implant standalone procedure versus classic trabeculectomy standalone procedure.

The primary endpoint is the proportion of patients with a best corrected distance visual acuity > 0.3 (logMAR) after 1 week.

Secondary objectives are the distance and near best corrected visual acuity measured at postoperative visits (e.g. day 1, month 1, 3, 12) and relative change of visual acuity at postoperative visits compared to baseline in both groups (e.g. month 1). The proportion of patients with a loss of best corrected distance visual acuity ≥ 2 lines at postoperative visits (e.g. day 1), the proportion of patients with a best corrected distance visual acuity (logMAR) > 0.3 and > 0.5 will be assessed at different postoperative visits (e.g. week 1, 2, month 1 and 3). Additionally, the time of recovery of visual acuity and the postoperative changes of refraction after the procedures will be compared. Secondary endpoints also include efficacy and safety of both procedures.

Subjects will undergo study visits at the following times: Preoperative Visit 1 (Screening), Operative Visit 2, 1 Day, 1 Week, 2 Weeks, 1 Month, 3, 6 Months, 12 Months Visit.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of open angle glaucoma (Primary open angle glaucoma, Pseudoexfoliation glaucoma, Pigmentary dispersion glaucoma)
2. Clinically eligible for both surgeries (Trabeculectomy and XEN) on the discretion of the surgeon (area of healthy, free and mobile conjunctiva in the superior nasal target quadrant)
3. VA logMAR ≤ 1 (VA dec ≥ 0.1)
4. Trabecular meshwork must be visible (with Shaffer angle grade > 1 in the target quadrant)
5. Age 18 years or older
6. Patient understands the nature of the procedure, is willing to comply with associated follow-up evaluations, and provides written informed consent

Exclusion Criteria:

1. Clinical significant cataract
2. Subject has had prior cataract surgery in study eye ≤ 1 months (count to operation)
3. Subject has had prior (incisional) glaucoma surgery (XEN, trabeculectomy, viscocanalostomy, canaloplasty, shunts of any type, collagen implants, etc.). Prior iridotomy is acceptable.
4. Phacic Angle Closure Glaucoma
5. Subject has neovascular, uveitic or angle recession glaucoma or any glaucoma associated with vascular disorders
6. Active inflammation (e.g., blepharitis, conjunctivitis, keratitis, uveitis)
7. Anterior chamber intraocular lens
8. Vitreous present in the anterior chamber
9. Presence of intraocular silicone oil
10. History of corneal surgery, corneal opacities, or corneal disease
11. Impaired episcleral venous drainage (e.g. Sturge-Weber or nanophthalmos)
12. History of dermatologic keloid formation
13. Active diabetic retinopathy, proliferative retinopathy, choroidal neovascularization, branch retinal vein occlusion, central retinal vein occlusion, or other ophthalmic disease or disorder that could confound study results
14. Known or suspected allergy or sensitivity to drugs required for the surgical procedure or any of the device components (e.g., porcine products or glutaraldehyde),
15. Pregnant or nursing women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Estimated)
Dates: Start 2023-12-20 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Best Corrected Distance Visual Acuity at 1 Week | Week 1
  The primary endpoint is the proportion of patients with a best corrected distance visual acuity > 0.3 (logMAR) after 1 week.

CONTACTS AND LOCATIONS:
Overall Officials: Herbert Reitsamer, MD, Study Chair — Paracelsus Medical University Salzburg/ Salzburger Landeskliniken
Locations (1):
- Dept. Ophthalmology and Optometry Paracelsus Medical University, Salzburg, Austria

IPD SHARING:
Plan to Share IPD: No